CLINICAL TRIAL: NCT01361542
Title: Effect Of Anti TNF Alpha Therapy On Disease Activity And Bone Health, And Their Adverse Effects In Ankylosing Spondylitis In A North Indian Population
Brief Title: Effect Of Anti TNF Alpha Therapy And Their Adverse Effects In Ankylosing Spondylitis In A North Indian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SKS/ASTNF/TB/2011
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Ankylosing Spondylitis
Keywords: TNF; BMD; Ankylosing spondylitis; bone health; Anti TNF therapy; Disease activity
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti TNF (Experimental): Anti TNF alpha therapy including either infliximab or etanercept with data obtained before and after the study duration.
  Interventions: Drug: anti TNF alpha agent; Drug: Anti TNF alpha therapy

INTERVENTIONS:
Drug: anti TNF alpha agent — Anti TNF alpha therapy included either INFLIXIMAB or ETANERCEPY Infliximab at 3-5 mg/kg at recommended protocols for the duration of the study Etanercept at 50mg weekly for the duration of the study
  Other Names: Infliximab - REMICADE as brand name; Etanercept- ENBREL as brand name
Drug: Anti TNF alpha therapy — Infliximab 3-5 mg/kg as per recommended protocol or Etanercept 50mg/week for 1 year
  Other Names: REMICADE-infliximab; ENBREL-Etanercept

SUMMARY:
Ankylosing Spondylitis (AS) is a chronic painful progressive inflammatory arthritis of unknown etiology primarily affecting the spine and sacroiliac joints. In addition to formation of new bone leading to syndesmophytes and ankylosis; osteoporosis is also a prominent feature in AS-thus showing the paradox of new bone formation at abnormal sites coexisting with reduced bone mass & increased fracture risk. Osteoporosis is a common complication of AS, with an incidence between 18.7% and 62%. TNF alpha has a central role in disturbing this balance in bone metabolism--resulting in accelerated alveolar bone loss and decreased strength- i.e. osteoporosis. The investigators hypothesis that anti TNF therapy is effective in active AS resistant to conventional therapy and helps in improving the bone density and over all bone health.

DETAILED DESCRIPTION:
Ankylosing spondylitis not responding to conventional therapy has been effectively treated with Anti TNF therapy. In addition studies have shown that TNF has a role in osteoporosis of inflammatory diseases. The hypothesis that anti TNF therapy may decrease osteoporosis and tilt bone metabolism to the osteoblastic side has been tested in few studies. These have not been studied in an Indian population. Another great issue in the usage of anti TNF therapy in Indian population is the high incidence of developing infective complications; especially tuberculosis. The investigators are thus studying these in a north Indian population at a tertiary centre. The results would come to important conclusions regarding treatment and in the important issue of tuberculosis screening and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are fulfilling the Modified New York Criteria(1984) for the diagnosis of Ankylosing Spondylitis
* Age ≥ 18 years
* Patients who have been planned to be started on anti Tnf alpha agents.
* Patients who have given consent for the study.

Exclusion Criteria:

* Patients with other coexistent rheumatologic diseases.
* Patients who have previously received anti TNF alpha agents in the past 1 year.
* Patients who are receiving other medications that may significantly alter the bone metabolism (like steroids, bisphosphonates, estrogen replacement therapy etc)
* Patients with any contraindications against the usage of anti TNF alpha agents (Active/ chronic infections, liver dysfunction, demyelinating diseases, pregnancy etc)
* Patients with other definite risk factors for osteoporosis like chronic alcoholism, smoking, endocrine disorders etc

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Increase in bone mineral density and decrease in disease activity | 2 years

SECONDARY OUTCOMES:
Observation of adverse effects of Anti TNF therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Franck H, Meurer T, Hofbauer LC. Evaluation of bone mineral density, hormones, biochemical markers of bone metabolism, and osteoprotegerin serum levels in patients with ankylosing spondylitis. J Rheumatol. 2004 Nov;31(11):2236-41. PMID 15517638